CLINICAL TRIAL: NCT05352984
Title: Risk Factors Assessment and Postponement Rate of Elective Surgical Procedures in Tertiary Care Public Sector Hospitals, Peshawar, Khyber Pakhtunkhwa, Pakistan-A Multicenter Cross-sectional Study
Brief Title: Postponement Rate of Elective Surgical Procedures
Acronym: Postponement
Status: Completed | Type: Observational
Sponsor: Hayatabad Medical Complex (Other Government)
Responsible Party: Principal Investigator, Rahman Ullah Jan, Principal investigator, Hayatabad Medical Complex
Other Study IDs: 616/HEC/B&PSC/2022
Record Dates: First submitted 2022-04-25; First posted 2022-04-29 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Surgical Procedure
Keywords: Postponement; Cancellation; Elective

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Postponement of elective surgical procedures is a major issue in health care facilities. It increases burden on hospitals and healthcare systems as well as misery of the patients and their family members. Patient's stay in the hospitals is prolonged. Hospitals and patients resources are wasted and their expenses are increased. The rate of postponement is different in different regions. It is estimated to be in between 9 to 44 %. Reason may be organizational or medical. Elective procedures are cancelled due to insufficient OT timings, non-availability of; anesthetists, blood or beds in ICU, change of plan and medical reasons like respiratory infections, cardiac problems, hypertension and uncontrolled diabetes. Tertiary care hospitals in Peshawar, Khyber Pakhtunkhwa, Pakistan are overburdened and patients on OT list are frequently postponed. Operating room timings has been increased to overcome the issue but no recent data is available regarding actual postponement rate and possible causes in this region. The need is felt to assess the problem and suggest recommendations to decrease patients' sufferings and improve hospital workings.

DETAILED DESCRIPTION:
Standardized surgical health care and its availability to every person in a community should the objective of a good health system but this is abstruse to complete especially in low and middle income countries. One reason for failure to complete this objective is postponement in elective surgical procedures. It increases burden on hospitals/ healthcare systems as well as misery of the patients and their family members. Patient's stay in the hospitals is prolonged. Hospitals and patients resources are wasted and their expenses are increased. Hospital resources like operation theatre (OT) are underutilized. Surgeons, nursing and other support staff's time is used worthlessly. Patients and attendants face economic and psychological stress. They bear extra financial burden due to stay in hospitals as well as leaves from work. They face more anxiety (42.1 %) and depressive disorders (26.3 %). Patient's health and outcome may deteriorate especially in cardiac, thoracic and cancer patients or in severe category or moribund patients waiting for their surgery.

Pakistan's health care system is based on public and private sector. Public sector health setups provides most facilities free of cost to the community. It is based on primary, secondary and tertiary health care setups. But they are not well integrated and proper referral system to secondary and tertiary health care is weak. Patients are unduly referred to tertiary care hospitals in more than their expected strengths by private clinics as well as by primary and secondary health care setups . Also because of our weak primary and secondary care system, patients coming to tertiary care setups are not aware of their comorbidities like Hypertension, diabetes, ischemic heart diseases, endocrine and respiratory diseases. We also receive fair number of referred patients from our neighboring country; Afghanistan. Some patients admitted for surgical procedures are postponed and are rescheduled for procedures in later dates, thus putting additional burden upon already overburdened system. The rate of postponement is different in different regions. It is estimated to be in between 9 to 44 %. Reason may be organizational or medical. Elective procedures are cancelled due to insufficient OT timings, non-availability of; anesthetists, blood or beds in ICU, change of plan and medical reasons like respiratory infections, cardiac problems, hypertension and uncontrolled diabetes. Cardiac surgeries, cancer surgeries, cholecystectomies, pediatric surgeries and thoracic surgeries are commonly postponed. In an older study done in 2007 in Abbotabad, Khyber Pakhtunkhwa, Pakistan, the postponement rate was 25 %. Elective procedures were cancelled due to shortage of time (36 %), beds (16.2 %), anesthetists (5.8 %) and medical reasons (31%) . Tertiary care hospitals in Peshawar, Khyber Pakhtunkhwa, Pakistan has increased the OR duration from 06 hours to 08 hours and so it is needed to know the new prevalence of cancellation rate of elective procedures and its causes adversely affecting the patients and hospital.

Rationale of the study: Tertiary care hospitals in Peshawar, Khyber Pakhtunkhwa are overburdened and patients on OT list are frequently postponed. Operating room timings has been increased but no recent data is available regarding actual postponement rate and possible causes in this region. The need is felt to assess the problem and suggest recommendations to decrease patients' sufferings and improve hospital workings.

Objectives: To assess the risk factors and postponement rate of elective surgical procedures on the same day of surgery in public sector tertiary care hospitals in Peshawar, Khyber Pakhtunkhwa, Pakistan.

Postponement is defined as cancellation of scheduled elective procedure on the day of operation.

ELIGIBILITY:
Inclusion Criteria:

* All inpatients of any age and either sex admitted in general surgery departments, scheduled for elective surgeries including laparoscopic surgeries, who arrive or are brought to operation theatre for general surgeries as elective cases.

Exclusion Criteria:

* All outdoor patients.
* Indoor cases of cardiac, cardiovascular, obstetrics and gynecology, neurosurgery, orthopedics, pediatrics or transplant surgeries or other surgeries considered as specialized surgeries.
* Emergency surgeries.

Min Age: 15 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All inpatients admitted in surgical departments of three tertiary care hospitals[ MTI-(HMC, KTH,LRH)], Peshawar, Pakistan and scheduled for elective general surgical procedures.
Sampling Method: Non-Probability Sample
Enrollment: 1221 (Actual)
Dates: Start 2022-05-19 (Actual); Primary Completion 2022-08-19 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
Postponement rate of elective surgical procedures | Eight hours
  Postponement/ cancellation rate of elective surgical procedures on the same day of surgery will be calculated.
  Postponement rate= Total number of elective procedures cancelled / Total number of general surgeries performed in the defined time period * 100

SECONDARY OUTCOMES:
Risk factors assessment of postponement | Eight hours
  Risk factors for postponement of elective surgical procedures on the same day of surgery will be assessed for presence or absence though a questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Rahman U Jan, Principal Investigator — Hayatabad Medical Complex
Locations (1):
- Hayatabad Medical Complex, Peshawar, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Data including clinical and demographic characteristics, not affecting patient's confidentiality, will be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: December, 2022 to December, 2025
Access Criteria: IPD will be shared on inter institutional request basis.

REFERENCES:
- [Background] Meara JG, Leather AJ, Hagander L, Alkire BC, Alonso N, Ameh EA, Bickler SW, Conteh L, Dare AJ, Davies J, Merisier ED, El-Halabi S, Farmer PE, Gawande A, Gillies R, Greenberg SL, Grimes CE, Gruen RL, Ismail EA, Kamara TB, Lavy C, Lundeg G, Mkandawire NC, Raykar NP, Riesel JN, Rodas E, Rose J, Roy N, Shrime MG, Sullivan R, Verguet S, Watters D, Weiser TG, Wilson IH, Yamey G, Yip W. Global Surgery 2030: evidence and solutions for achieving health, welfare, and economic development. Lancet. 2015 Aug 8;386(9993):569-624. doi: 10.1016/S0140-6736(15)60160-X. Epub 2015 Apr 26. No abstract available. PMID 25924834
- [Background] Abate SM, Chekole YA, Minaye SY, Basu B. Global prevalence and reasons for case cancellation on the intended day of surgery: A systematic review and meta-analysis. Int J Surg Open. 2020;26:55-63. doi: 10.1016/j.ijso.2020.08.006. Epub 2020 Aug 20. PMID 34568611
- [Background] O'Rielly C, Ng-Kamstra J, Kania-Richmond A, Dort J, White J, Robert J, Brindle M, Sauro K. Surgery and COVID-19: a rapid scoping review of the impact of the first wave of COVID-19 on surgical services. BMJ Open. 2021 Jun 15;11(6):e043966. doi: 10.1136/bmjopen-2020-043966. PMID 34130956
- [Background] Tagarakis GI, Voucharas C, Simopoulos V, Karangelis D, Daskalopoulos ME, Parisis C, Tsantilas A, Sataitidis I, Lampoura S, Vretzakis G, Tsilimingas NB. Why are thoracic operations postponed? J Cardiothorac Surg. 2012 Apr 11;7:31. doi: 10.1186/1749-8090-7-31. PMID 22494485
- [Background] Kurji Z, Premani ZS, Mithani Y. Analysis Of The Health Care System Of Pakistan: Lessons Learnt And Way Forward. J Ayub Med Coll Abbottabad. 2016 Jul-Sep;28(3):601-604. PMID 28712245
- [Background] Sommer JL, Jacobsohn E, El-Gabalawy R. Impacts of elective surgical cancellations and postponements in Canada. Can J Anaesth. 2021 Mar;68(3):315-323. doi: 10.1007/s12630-020-01824-z. Epub 2020 Oct 21. PMID 33085061
- [Background] marymarcus. CAUSES OF POSTPONEMENT OF ELECTIVE SURGERY IN MAYO HOSPITAL LAHORE [PDF] [Internet]. Presentica. 2020 [cited 2021 Dec 27]. Available from: https://www.presentica.com/doc/10371391/causes-of-postponement-of-elective-surgery-in-mayo-hospital-lahore
- [Background] Bathla S, Mohta A, Gupta A, Kamal G. Cancellation of elective cases in pediatric surgery: An audit. J Indian Assoc Pediatr Surg. 2010 Jul;15(3):90-2. doi: 10.4103/0971-9261.71748. PMID 21124662
- [Background] Zafar A, Mufti TS, Griffin S, Ahmed S, Ansari JA. Cancelled elective general surgical operations in Ayub Teaching Hospital. J Ayub Med Coll Abbottabad. 2007 Jul-Sep;19(3):64-6. PMID 18444594